CLINICAL TRIAL: NCT02477124
Title: A See and Treat Paradigm for Cervical Pre-cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00052865
Record Dates: First submitted 2015-06-12; First posted 2015-06-22 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cervical Pre-cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- transvaginal digital colposcope (TVCD) (Active Comparator): Each enrolled patient will undergo the standard of care for cervical cancer screening at her institution, and then the trans-vaginal colposcope will be used to collect digital images of the cervix.
  Interventions: Device: transvaginal digital colposcope (TVDC)
- standard of care screening (Active Comparator): Each enrolled patient will undergo the standard of care for cervical cancer screening at her institution, and then the trans-vaginal colposcope will be used to collect digital images of the cervix.
  Interventions: Other: Standard of care screening

INTERVENTIONS:
Device: transvaginal digital colposcope (TVDC) — TVDC is a miniature colposcope used to obtain images of cervical tissue.
  Arms: transvaginal digital colposcope (TVCD)
Other: Standard of care screening — Standard of care screening varies from institution to institution but is either visual inspection with the naked eye, colposcopy, or visual inspection with a camera or microscope
  Arms: standard of care screening

SUMMARY:
The purpose of this study is to see if the transvaginal colposcope produces similar results to colposcopy for the screening of cervical cancer. In this study the investigators are using an investigational device called the transvaginal colposcope. The word investigational means that the device is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cervicography OR colposcopy OR VIA OR patients undergoing LEEP for the treatment of cervical cancer.
* Age 25 and greater
* Patients of all ethnic backgrounds will be included.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Children and subjects under 25.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2015-09; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala Ramanujam, PhD, Principal Investigator — Duke University
Locations (5):
- Duke University Medical Center, Durham, North Carolina, United States
- AIIMS, New Delhi, India
- La Liga Contra el Cancer, Lima, Peru
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania
- University Teaching Hospital, Lusaka, Zambia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cervical images obtained across 6 countries to build a database of 1000+ images to develop AI software for cervical cancer screening.
Period: Overall Study
Arm/Group | Transvaginal Digital Colposcope (TVCD)
Started | 514
Completed | 514
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transvaginal Digital Colposcope (TVCD)
Number analyzed (Participants) | 514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 514
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 200
  Not Hispanic or Latino | 314
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 125
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 189
  White | 200
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 100
  Zambia | 89
  Peru | 200
  India | 125

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which the Standard of Care Diagnosis and the Diagnosis of the TVDC Image Agree
Time Frame: Up to approximately 10 minutes
Population: We have SOC Images from these 514 participants AND the images obtained with our research device. Therefore we have 2 photos for each step in the colposcopy procedure process
Measure: Count of Participants; unit: Participants
Arm/Group | Transvaginal Digital Colposcope (TVCD)
Number analyzed (Participants) | 514
Participants | 514

ADVERSE EVENTS:
Time Frame: Until pathology results are available, up to approximately 14 days
Arm/Group | Transvaginal Digital Colposcope (TVCD)
All-Cause Mortality (participants affected / at risk) | 0/514
Serious Adverse Events (participants affected / at risk) | 0/514
Other Adverse Events (participants affected / at risk) | 0/514

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02477124/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02477124/ICF_001.pdf